CLINICAL TRIAL: NCT04652219
Title: Clinical Study on the Safety and Efficacy of CART Cells in the Treatment of Advanced GUCY2C-positive Digestive Tract Tumors
Brief Title: CART Therapy in GUCY2C-positive Digestive Tract Tumors
Acronym: CART
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Weijia Fang, MD (Other)
Collaborators: Innovative Cellular Therapeutics Co., Ltd. (Other)
Responsible Party: Sponsor-Investigator, Weijia Fang, MD, director, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-GC
Record Dates: First submitted 2020-11-09; First posted 2020-12-03 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Malignant Neoplasms of Digestive Organs
Keywords: cart; gucy2c; Digestive tract tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with late malignant digestive tract tumor (Experimental): Patients with late malignant digestive tract tumor, for example metastatic colorectal cancer, pancreatic cancer, gastric cancer and so on. because of this is a open, single arm trail, there is no control group.
  Interventions: Biological: gucy2c cart cells

INTERVENTIONS:
Biological: gucy2c cart cells — Patients with advanced malignant gastrointestinal tumors were injected with CART cells

SUMMARY:
Ict-gc is an open, single-center study to evaluate the safety and efficacy of CAR-T-targeted therapy in patients with advanced gastrointestinal tumors.

DETAILED DESCRIPTION:
The primary objective of phase 1 is to evaluate the safety of CART regimens. The primary objective of phase 2 is to evaluate the efficacy of CART, as measured by objective response rate in subjects with colorectal cancer. Secondary objectives will include assessing the safety and tolerability of CART and additional efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70; 2. Positive expression of immunohistochemical (IHC) assay targets in a laboratory approved by the partner; 3. Pathology confirmed digestive tract tumor; 4. Patients who have failed or relapsed after at least the first and second line standard treatment, and patients who are intolerant to or voluntarily give up the standardized treatment; 5. At least one extracranial measurable lesion according to RECIST1.1 or EORTC or PERCIST; 6. Expected survival ≥90 days; 7. The main organs are functioning normally, i.e. they meet the following criteria:

1. ECOG physical condition score is 0~1 or KPS score is >70;
2. serum test criteria were as follows: HB≥90g/L (no blood transfusion within 14 days), ANC≥ 1.5 x 10^9/L, PLT≥80 x 10^9/L, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×ULN (upper limit of normal value).
3. Biochemical examination shall meet the following standards: TBIL≤ 1.5x ULN (upper limit of normal value); ALT and AST≤ 2.5x ULN; ALT and AST≤5xULN in case of liver metastasis; Serum Cr≤1xULN, endogenous creatinine clearance rate >50 ml/min (Cockcroft-Gault formula);
4. cardiac ejection fraction >55%; 8. No hemorrhagic disease or coagulation disorder; 9. No allergy to the developer; 10. Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days prior to enrollment, with negative results, and be willing to use an appropriate method of contraception during and 8 weeks after the last dose of CART (women who have undergone sterilization or have been postmenopausal for at least 2 years may be considered sterile); 11. The subjects voluntarily joined the study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. T cell transduction efficiency <5% or T cell amplification < 2 times after culture;
2. Participated in other drug clinical trials within 4 weeks before the start of the study;
3. Patients with hypertension and unable to obtain good control by single antihypertensive drugs (systolic blood pressure > 140 mmHg, diastolic blood pressure b> 90 mmHg, the specific conditions shall be evaluated by the researchers) have myocardial ischemia or infarction of grade I or above, arrhythmia of grade I or above (including QT interval ≥ 440ms) or cardiac insufficiency;
4. A wound or fracture in the chest or other area that has not healed for a long time;
5. Has a history of substance abuse and is unable to quit or has a history of mental disorders;
6. Patients with past or present objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, severe pulmonary function impairment, etc.;
7. Fungus, bacteria, virus or other infection that cannot be controlled or requires antibiotic treatment. The presence of a simple urinary tract infection and uncomplicated bacterial pharyngitis is permitted after consultation with a medical supervisor;
8. For subjects who have used chemotherapy before, according to NCI-CTCAE 4.0, there is grade ≥2 hematological toxicity or grade ≥3 non-hematological toxicity at the time of enrollment;
9. A known history of HIV, or a positive nucleic acid test for hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive);
10. The presence of any indwered catheter or drainage tube (e.g., bile drainage tube or pleural/peritoneal/pericardial catheter). The use of specialized central venous catheters was permitted (the influence of fistula, percutaneous nephrostomy, and indwsed Foley catheters in colorectal cancer patients was considered by the investigators);
11. Brain metastases; A history or medical condition of CNS, such as seizure disorder, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving CNS;

13. Significant immunodeficiency; 14. The major therapeutic drugs in this study (including fludalabine, cyclophosphamide, sodium meth, and tozumab and anti-infective drugs used to prevent and treat CRS) have a history of severe hypersensitivity reaction; 15. History of deep vein thrombosis or pulmonary embolism 6 months before enrollment; 16. A history of an autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) that has resulted in injury to the terminal organs or that requires systemic immunosuppressive/disease-modulating drugs in the past 2 years; 17. Any disease that may interfere with the evaluation of the safety or efficacy of the study treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2021-10-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with CAR-T treatment-related adverse events as assessed by CTCAE v4.03 | 24 months
  The investigator is responsible for ensuring that all adverse events observed by the investigator or reported by the subject during the 3-month period from enrollment (i.e. initiation of leukocyte separation) to 3 months after targeted car-t infusion are monitored and reported. After three months, researchers will be required to monitor and report targeted adverse events, including neurological, blood, infection, autoimmune diseases, and secondary malignant tumors, for 24 months or until disease progression, whichever occurs first.

SECONDARY OUTCOMES:
The event of cytokine release syndrome was reported using the grading scale in the protocol. | 24 months
  We will summarize the classification of cytokine release syndrome (CRS) according to the severity and system organ classification.
Efficacy will be assessed according to RECIST1.1 or EORTC or PERCIST criteria. | 24 months
  Remission will be evaluated by the central investigator at the time indicated in the evaluation plan. The disease was evaluated according to the response evaluation criteria in solid tumors RECIST version 1.1 or EORTC or percist. Flow cytometry, molecular or cytogenetic studies used in the trial will be used to assist, but will not be used alone to determine remission.

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, Principal Investigator — First Affiliated Hospital,Zhejiang University
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No